CLINICAL TRIAL: NCT05190536
Title: Ho:YAG Laser Versus Thulium Laser for the Management of 2-4cm Kidney Stones During SMP（Suction Mini Percutaneous Nephrolithotomy）：An International Multicenter Randomized Controlled Trial
Brief Title: Ho:YAG Laser Versus Thulium Laser for the Management of 2-4cm Kidney Stones During SMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMU Multicentre RCT2022
Record Dates: First submitted 2022-01-04; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Kidney Stones
Keywords: SMP; Ho:YAG; TFL; Kidney calculi; Efficency; Safety
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Patients in Group 1 undergo Ho:YAG laser (Experimental)
  Interventions: Procedure: Ho:YAG lasers
- Experimental: Patients in Group 2 undergo TFL (Experimental)
  Interventions: Procedure: TFL

INTERVENTIONS:
Procedure: Ho:YAG lasers — Under the guidance of B-ultrasound or X-ray, the appropriate target calyx was punctured with an 18G puncture needle.Percutaneous tract was established with 18Fr suction sheath. 12Fr nephroscope and 360um Ho:YAG laser fiber was used for lithotripsy.Kidney stones were fragmented by Ho:YAG lasers, and sucked out by the suction sheath.
  Arms: Experimental: Patients in Group 1 undergo Ho:YAG laser
Procedure: TFL — Under the guidance of B-ultrasound or X-ray, the appropriate target calyx was punctured with an 18G puncture needle.Percutaneous tract was established with 18Fr suction sheath. 12Fr nephroscope and 360um TFL fiber was used for lithotripsy.Kidney stones were fragmented by TFL, and sucked out by the suction sheath.
  Arms: Experimental: Patients in Group 2 undergo TFL

SUMMARY:
With the rapid development of medical equipment and the increasing experience, minimally invasive percutaneous nephrolithotomy (mini-PCNL) has been a well established modality for the management of upper urinary tract stones. The introduction of negative pressure suction technology into mini-PCNL can actively suck out the perfusion fluid and stone fragments, therefore to speed up stone removal efficency and keep a low intrarenal pressure, and was called suction mini-PCNL (SMP).

The common energy sources for SMP were pneumatic ballistic lithotripsy and Ho:YAG laser. The handle of pneumatic ballistic lithotripsy was heavy and can not be fixed on the nephroscope, furthermore, the fragments in pneumatic ballistic lithotripsy was large, therefore the active suction and discharge of stone fragments can not be well completed at the same time of lithotripsy. However, the Ho:YAG laser can well match the requirement of SMP that lithotripsy and suction can work at the same time. Recently, thulium fiber laser (TFL) was also used for lithotripsy. The versatility of TFL, including high frequencies and reduced retropulsion may result in higher ablation efficiency compared to Ho:YAG laser. However, there is no clinical study on the difference between Ho:YAG laser and thulium laser in SMP, which limits the reasonable choice of laser in SMP to a certain extent.

So, the investigators would like to have an international multi-centre RCT to compare the therapeutic effects of SMP with Ho:YAG laser versus TFL in the treatment of 2-4cm renal calculi, so as to provide high-level evidence to support for clinical selection.

DETAILED DESCRIPTION:
To compare the therapeutic effects of SMP with Ho:YAG laser versus TFL in the treatment of 2-4cm renal calculi，an international multi-centre RCT was conducted with the comparision of Ho:YAG laser and Thulium laser . Investigators plan to do an international multi-centre randomized controlled trial (RCT).

There are 20 hospitals from China, USA, United Kingdom, Italy, Spain, Sweden, Kuwait, Turkey, Philippines, Bulgaria and others.

The primary study endpoints was operation time,while the secondary study endpoints were stone free rate (SFR), postoperative hemoglobin drop, blood transfusion, postoperative fever and other complications.

This study will be started at March，2022 and ended at December,2024.

According to the literature and unpublished data from clinical practice or trails, the operative time of SMP with Ho:YAG laser and TFL for treating 2-4cm kidney stones was about 50±10.0 and 60±10min. It was assumed that the operation time of SMP using TFL was longer than that of SMP using Ho:YAG laser, the test level Type-1 error (α) was 0.05, the test efficiency power (1-β) was 0.8, the ratio of the two groups of sample size was 1:1, the non-inferiority test threshold was -12, and 310 was calculated for each group. Taking into account disengagement and other problems, n=341 was required in each group, therefore a total of 682 cases were required in the present RCT.

In the present study, the balanced random method was used to generate a random number table and randomly assign patients to each group. Considering the time zone difference of each country, the randomization cannot be arranged in real time, so the central randomized allocation method was adopted, package with certain cases and initial randomization was sent to the sub center, so as to ensure that there will be no excessive deviation in the number of cases completed by each sub center.

Patients received standard preoperative evaluation, including detailed medical history, physical examination, compete blood count, urinary analysis, midstream urine culture, serum creatinine, electrolyte biochemical tests, coagulation profiles, blood-borne disease screening, non-contrast CT, plain radiography (kidney ureter bladder, KUB), plain chest radiograph, electrocardiogram etc.

The number of annual SMP operations required for inclusion center was≥200, and the main researchers carried out SMP was≥50 each year. Both laser were required in the hospital.

Patients received standard preoperative evaluation, including detailed medical history and examination. On the 1 day before operation, the eligible patients were arranged according to the random number that have been generated to the group, "0" for Ho:YAG laser group, while "1" for TFL group.

All procedures were under general anesthesia. Firstly, in lithotomy position, 5Fr ureteral catheter was retrogradely placed into the affected ureter, and the patient was transferred to prone position.Under the guidance of B-ultrasound or X-ray, the appropriate target calyx was punctured with an 18G puncture needle. The fascial dilator was used to dilate the tract to 18Fr, and percutaneous tract was established with 18Fr suction sheath. 12Fr nephroscope and 360um laser fiber was used for lithotripsy. Kidney stones were fragmented by lasers, and sucked out by the suction sheath. At the later stage of the procedure, fluoroscopy was performed to detect the residual stone. Further attempt was made to remove all stone. Double-J stent and/or nephrostomy tube was inserted. Tubeless PCNL was feasible if there was no residual stones, no bleeding, no collecting system perforation nor no ureteral obstruction.

All the stone fragments was collected and the volume of removing stones was evaluated、Stone compositon analysis was obtained for all patient.Complete blood count and electrolyte biochemical tests were performed at 8:00 the next morning after surgery. KUB was required on the 2nd postoperative day to evaluate the stone, stent, and tube status.If the stones were completely removed with no additional procedures needed, the patient is discharged after removing nephrostomy tube .If the residual fragments are≧4mm, any information concerning needs for auxiliary treatment（RIRS、PCNL、SWL） will be recorded, including the size of the residual stone, the method of adjuvant therapy and the final outcomes.Two weeks after surgery, the final SFR was determined by KUB and the JJ stent was removed.

Data collection and definitions of parameters The characteristics of patients and clinical outcomes were recorded according to the pre-established case report form (CRF). Surgical outcomes were predicted preoperatively according to the S·T·O·N·E nephrolithometry. Puncture guidance#Sonography/X ray/ combination#, tract location#lower, middle, upper pole and supracostal or subracostal#, tract number, lithotripsy tool, tube and setnt (nephrostomy tube, JJ stent or tubeless). Operation time was defined as the time from puncture to the placement of the nephrostomy tube. Lithotripsy time was defined as the time for lithotripsy only. Hospital stay was defined as days between the surgery date and discharge date. Bruggrmann Comfort Scale (range: 0-5): 0, persistent pain; 1, severe pain while deep breathing or coughing; 2, mild pain while deep breathing or coughing; 3, no pain while deep breathing; 4, no pain while coughing. (Ren C et al. Medicine (Baltimore). 2015 Aug;94(32):e1348.). Visual Analogue Scale (range: 1-10): 0, no pain; 1-3, mild; 4-6, moderate; 7-9, severe; 10, excruciating pain. (Reed MD, Van Nostran W. J Clin Pharmacol. 2014 Mar;54(3):241-4.). Postoperative fever was defined as armpit temperature≥38#. SIRS was diagnosed in patients who met two or more of the following clinical findings: # body temperature higher than 38# or lower than 36#;# heart rate higher than 90 beats per minute; # respiratory rate greater than 20 breaths per minute or PaCO2 less than 32mm Hg; # a white blood cell count higher than 12,000 per mm 3 or lower than 4,000 per mm3. Urosepsis was diagnosed with SOFA scores. Complications of all patients were recorded according to modified Clavien classification system.

Statistical Package for Social Sciences (SPSS) 22.0 was used for statistical analysis. Continuous data were recorded as mean ± standard deviation. Normally distributed data were analyzed with Student's t test, while non-normally distributed data were analyzed with Mann-Whitney U test. Categorical data were reported as n (%), and compared with the χ2 test or Wilcoxon rank sum test. p < 0.05 was regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. 2-4cm kidney stones.
2. Aged 18-70 years.
3. SMP with Ho:YAG laser or TFL.

Exclusion Criteria:

1. Transplanted kidney, solitary kidney, horseshoe kidney, urinary diversion, urethra deformity and other special cases.
2. If empyema was found during SMP, the nephrostomy tube was retained and the patient was excluded from the trail.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Operation time | Intraoperative (the time from puncture to the placement of the nephrostomy tube)
  Operation time is defined as the time from puncture to the placement of the nephrostomy tube

SECONDARY OUTCOMES:
Stone free rate (SFR) | 1 month after removing the pigtail stent
  2mm Non-contrast CT is obtained for all patients at one month after removing the pigtail stent to evaluate the final SFR. Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were definded as ≤ 4mm, asymptomatic, non-obstructive and non-infectious stone particles
postoperative fever | ≤ 1month postoperatively
  Postoperative fever was defined as armpit temperature ≥38C
Complications is defined as any adverse event occurred | intraoperatively or ≤ 1month postoperatively
  Complications is defined as any adverse event occurred intraoperatively or ≤ 1month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, Ph.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong,China, China

REFERENCES:
- [Background] Becker B, Gross AJ, Netsch C. Ho: YaG laser lithotripsy: recent innovations. Curr Opin Urol. 2019 Mar;29(2):103-107. doi: 10.1097/MOU.0000000000000573. PMID 30407221